CLINICAL TRIAL: NCT02991976
Title: Effects of High Inspiratory Oxygen on Cerebral Tissue Oxygenation and Patient Recovery After Carotid Endarterectomy
Brief Title: Oxygen Concentration and Recovery After Carotid Endarterectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Osijek University Hospital (Other)
Responsible Party: Principal Investigator, Vedran Gašić, MD, Vedran Gasic, M.D., Osijek University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: OsijekUH4
Record Dates: First submitted 2016-12-05; First posted 2016-12-14 (Estimated); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Hypoxia-Ischemia, Brain; Ischemia, Vertebral Artery; Artery Stenosis, Carotid
Keywords: Normobaric hyperoxia; Cerebral oxygenation; Near-infrared spectroscopy; Carotid endarterectomy; TIVA
MeSH Terms: conditions — Hypoxia-Ischemia, Brain; Vertebrobasilar Insufficiency; Carotid Stenosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 35% O2 (Active Comparator): Patient receiving 35% O2 during carotid endarterectomy, Intervention - oxygen concentration
  Interventions: Procedure: Oxygen concentration
- 100% O2 (Active Comparator): Patient receiving 100% O2 during carotid endarterectomy, Intervention - oxygen concentration
  Interventions: Procedure: Oxygen concentration

INTERVENTIONS:
Procedure: Oxygen concentration — Shunting, raising concentration of O2 because of improving regional cerebral oxygen saturation (rSO2), keeping blood pressure above 120-130 mmHg, positive end expiratory pressure (PEEP)

SUMMARY:
This study evaluates effects of high inspiratory oxygen on cerebral tissue oxygenation and patient recovery after carotid endarterectomy. Two group of patient undergoing to carotid with total intravenous anaesthesia will receive either 35% inspired oxygen or 100% oxygen.

DETAILED DESCRIPTION:
High inspired oxygen concentration may reduce brain hypoxia in the patients undergoing carotid endarterectomy with total intravenous anaesthesia. However, there are some studies suggesting that high inspired oxygen concentration may induce cerebral vasoconstriction. This study was performed to measure the influence of fraction of inspired oxygen (FiO2) on the regional tissue oxygenation in the patients undergoing carotid endarterectomy with total intravenous anaesthesia. The INVOS 5100B monitor was used for regional cerebral oxygen saturation (rSO2) measurement from operative and nonoperative side, and INVOS Analytics Tool (Covidien) for area under curve (AUC) calculations. A bispectral index and invasive blood pressure monitoring were used in all patients.

ELIGIBILITY:
Inclusion Criteria:

* patient undergoing surgery (carotid endarterectomy)

Exclusion Criteria:

* decompensated and uncontrolled respiratory and cardiac disease, myocardial infarction suffered in the last 6 months, cerebrovascular infarction, coagulopathy, anaphylaxis to drugs

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-11; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Area under curve of regional cerebral oxygen saturation (rSO2) curve | During surgery
  Intraoperative high oxygen concentrations may reduce intensity of tissue hypoxic episodes during carotid endarterectomy in total intravenous anesthesia (TIVA).
  The INVOS 5100B monitor was used for regional cerebral oxygen saturation (rSO2) measurement from operative and nonoperative side, and INVOS Analytics Tool (Covidien) for Area under curve (AUC) calculations. Data were analyzed using two sided T-test and Fisher exact test. A P<0.05 was considered as statistically significant Postoperative follow up in large patient's group is necessary to confirm its impact on patients' outcome.

SECONDARY OUTCOMES:
Early neurologic recovery, TIA or brain ischemia | Till 7 days after surgery
  Postoperative patient follow up by clinical signs or CT scan confirmation
Intensive Care Unit admission, Death | Till 7 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: slavica kvolik, prof., Study Director — Osijek Hospital University
Locations (1):
- Osijek Hospital University, Osijek, County of Osijek-Baranja, Croatia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rockswold SB, Rockswold GL, Zaun DA, Liu J. A prospective, randomized Phase II clinical trial to evaluate the effect of combined hyperbaric and normobaric hyperoxia on cerebral metabolism, intracranial pressure, oxygen toxicity, and clinical outcome in severe traumatic brain injury. J Neurosurg. 2013 Jun;118(6):1317-28. doi: 10.3171/2013.2.JNS121468. Epub 2013 Mar 19. PMID 23510092
- [Result] Picton P, Chambers J, Shanks A, Dorje P. The influence of inspired oxygen fraction and end-tidal carbon dioxide on post-cross-clamp cerebral oxygenation during carotid endarterectomy under general anesthesia. Anesth Analg. 2010 Feb 1;110(2):581-7. doi: 10.1213/ANE.0b013e3181c5f160. Epub 2009 Dec 2. PMID 19955500
- [Result] Nielsen HB. Systematic review of near-infrared spectroscopy determined cerebral oxygenation during non-cardiac surgery. Front Physiol. 2014 Mar 17;5:93. doi: 10.3389/fphys.2014.00093. eCollection 2014. PMID 24672486
- [Result] Rokamp KZ, Secher NH, Eiberg J, Lonn L, Nielsen HB. O2 supplementation to secure the near-infrared spectroscopy determined brain and muscle oxygenation in vascular surgical patients: a presentation of 100 cases. Front Physiol. 2014 Feb 25;5:66. doi: 10.3389/fphys.2014.00066. eCollection 2014. PMID 24611051
- [Result] Hojlund J, Sandmand M, Sonne M, Mantoni T, Jorgensen HL, Belhage B, van Lieshout JJ, Pott FC. Effect of head rotation on cerebral blood velocity in the prone position. Anesthesiol Res Pract. 2012;2012:647258. doi: 10.1155/2012/647258. Epub 2012 Sep 5. PMID 22988456
- [Result] Wolff CB. Oxygen delivery: the principal role of the circulation. Adv Exp Med Biol. 2013;789:37-42. doi: 10.1007/978-1-4614-7411-1_6. PMID 23852474